CLINICAL TRIAL: NCT01802502
Title: Explorative PK Study Comparing 600 mg Rifampicin i.v. With 750 mg and 900 mg Rifampicin Oral in Tuberculous Meningitis Patients
Brief Title: Rifampicin Explorative PK Study for Tuberculous Meningitis Comparing Oral and Intravenous Preparation
Acronym: REMOVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB-201302.01
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Tuberculous Meningitis
Keywords: tuberculous meningitis; rifampicin; bioequivalence; oral administration; intravenous administration
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rifampicin 600 mg (Active Comparator): Subjects in this arm receive 600 mg rifampicin intravenously
  Interventions: Drug: Rifampicin intravenous
- rifampicin 750 mg (Experimental): Subjects in this arm receive 750 mg rifampicin orally
  Interventions: Drug: Oral rifampicin
- rifampicin 900 mg (Experimental): Subjects in this arm receive rifampicin 900 mg orally
  Interventions: Drug: Oral rifampicin

INTERVENTIONS:
Drug: Rifampicin intravenous
  Other Names: Rifadin
  Arms: Rifampicin 600 mg
Drug: Oral rifampicin
  Other Names: Rifampisin (Kimia Farma, Bandung, Indonesia)
  Arms: rifampicin 750 mg; rifampicin 900 mg

SUMMARY:
Tuberculous (TB) meningitis is the most severe manifestation of TB infection, leaving up to 50% of patients dead or neurologically disabled. Current treatment is similar to treatment of lung TB, although penetration of some antibiotics into the brain is poor and the immune-pathology of TB meningitis is very different from pulmonary TB. In a recent phase II clinical trial from the investigators group, the first of its kind globally, intensified antibiotic treatment, with moxifloxacin and high dose rifampicin, strongly reduced mortality of TB meningitis.

The investigators aim to examine the effect of intensified antibiotic treatment on mortality and morbidity of TB meningitis in a phase 3 clinical trial, preceded with an explorative pharmacokinetic (PK) study to examine if higher oral doses rifampicin result in exposures similar to the i.v. dose used in our phase 2 trial, since oral rifampicin could be implemented much easier in low-resource settings.

DETAILED DESCRIPTION:
Introduction:

In a recent clinical trial the investigators have shown that a higher dose of rifampicin administered intravenously (600 mg iv) during the first 2 weeks of treatment is safe and associated with a survival benefit in adults with TB meningitis. An oral (rather than iv) dose would help implementation of intensified treatment for TB meningitis. However, it is hard to predict what oral dose of rifampicin will result in rifampicin exposures similar to 600 mg iv, due to differences in bio-availability (oral vs. iv) and the unpredictable dose-concentration relationship (nonlinear pharmacokinetics of rifampicin). Therefore the investigators aim to examine the pharmacokinetic of 2 higher doses of rifampicin (750 mg and 900 mg) given orally, and compare the pharmacokinetic profiles with the result of our previous study using 600 mg rifampicin iv.

General Objective:

To help establish the optimized treatment regimen for TB meningitis

Specific Objectives:

1. To explore whether exposures resulting from oral rifampicin 750 mg or 900 mg are similar to exposures after intravenous rifampicin 600 mg during the first two days of treatment
2. To explore whether exposures resulting from oral rifampicin 750 mg or 900 mg are similar to exposures after 14 days of treatment (stabilized rifampicin concentrations, i..e steady-state)
3. To evaluate the safety and tolerability of high dose of oral rifampicin
4. To evaluate neurological response and mortality after 2 weeks of treatment with high dose rifampicin

Study Design:

Explorative pharmacokinetic study; randomized, three-arm, two-period evaluation.

Study procedure:

After diagnosis of TB meningitis, eligible patients will be randomized to get either oral 750 mg, oral 900 mg, or iv 600 mg rifampicin for 14 days in combination with standard oral TB drugs (isoniazid 300 mg/day, ethambutol 750 mg/day, and pyrazinamide 1500mg/day) and adjuvant dexamethasone i.v. and pyridoxine.

Serial blood samples will be taken 6 times from 0, 1, 2, 4, 8, and 12 hour after drug administration at the first or second day of treatment and at day 14 (steady-state). Single cerebrospinal fluid (CSF) sample will be taken 3-6 hours after administration at the same day of blood sampling days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Probable/possible tuberculosis meningitis using uniform case definition
* Agree to participate in the study

Exclusion Criteria:

* Patient with antituberculosis treatment within last 2 weeks.
* Increase liver function >5x upper limit of normal
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of several rifampicin dose | Day 2 and Day 14; 6 time points for blood analysis, and 1 time point for CSF analysis
  We will measure plasma drug concentration at hour 0, 1, 2, 4, 8, and 12, while CSF drug concentration will be measured at a single time point i.e. at hour 3-6 post dose. The sampling days will be (1) within the first three days, and (2) at day 14 of the intensified treatment.

SECONDARY OUTCOMES:
mortality | early (1 month) and late (6 months)
  We will measure early and late mortality

CONTACTS AND LOCATIONS:
Overall Officials: Rovina Ruslami, M.D., PhD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran - Dr. Hasan Sadikin Hospital Bandung
Locations (1):
- Hasan Sadikin Hospital, Bandung, West Java, Indonesia

REFERENCES:
- [Background] Ruslami R, Ganiem AR, Dian S, Apriani L, Achmad TH, van der Ven AJ, Borm G, Aarnoutse RE, van Crevel R. Intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis: an open-label, randomised controlled phase 2 trial. Lancet Infect Dis. 2013 Jan;13(1):27-35. doi: 10.1016/S1473-3099(12)70264-5. Epub 2012 Oct 25. PMID 23103177
- [Background] Marais S, Thwaites G, Schoeman JF, Torok ME, Misra UK, Prasad K, Donald PR, Wilkinson RJ, Marais BJ. Tuberculous meningitis: a uniform case definition for use in clinical research. Lancet Infect Dis. 2010 Nov;10(11):803-12. doi: 10.1016/S1473-3099(10)70138-9. Epub 2010 Sep 6. PMID 20822958